CLINICAL TRIAL: NCT02916290
Title: Fuzhenghuayu in Combination With Ursodeoxycholic Acid in Primary Biliary Cirrhosis
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xijing Hospital of Digestive Diseases (Other)
Responsible Party: Principal Investigator, Han Ying, Professor Consultant Physician, Xijing Hospital of Digestive Diseases
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KY20151230-6
Record Dates: First submitted 2016-01-28; First posted 2016-09-27 (Estimated); Last update posted 2016-09-27 (Estimated); Status verified 2016-09

CONDITIONS: Primary Biliary Cirrhosis
Keywords: Fuzhenghuayu
MeSH Terms: conditions — Liver Cirrhosis, Biliary

ARMS (2):
- Fuzhenghuayu+UDCA (Experimental): Regular UDCA treatment combination with Fuzhenghuayu
  Interventions: Drug: Fuzhenghuayu; Drug: UDCA
- Monotherapy (Active Comparator): UDCA monotherapy
  Interventions: Drug: UDCA

INTERVENTIONS:
Drug: Fuzhenghuayu
  Arms: Fuzhenghuayu+UDCA
Drug: UDCA

SUMMARY:
Ursodeoxycholic acid (UDCA) has been the only treatment for PBC approved by US and European drug administrations. Long-term use of UDCA (13-15 mg/kg/day) in patients with PBC improves serum liver biochemistries and survival free of liver transplantation.

However, about 40% of patients do not respond to UDCA optimally as assessed by known criteria for biochemical response. Those patients represent the group in need for additional therapies, having increased risk of disease progression and decreased survival free of liver transplantation. And UDCA has less effect on PBC patients whose pathology stage 3-4. Liver fibrosis might jeopardize the UDCA effect. Fuzhenghuayu is a Chinese traditional medicine for liver fibrosis and cirrhosis. Both lab research and some clinical studies suggest that Fuzhenghuayu could significantly reverse liver fibrosis and cirrhosis due to different kind of etiology. Here the investigators start a random, open and parallel clinical research to explore the effect of Fuzhenghuayu combined with UDCA in the PBC treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent
2. Patient with PBC defined by 2 in 3 of the following criteria:

   * Positive antimitochondrial antibody type M2;
   * Abnormal serum alkaline phosphatases (ALP > 1,5N) and aminotransferase (AST or ALT > 1N) activities;
   * Histological hepatic injuries consistent with PBC.

Exclusion Criteria:

1. Pregnancy or desire of pregnancy.
2. Breast-feeding.
3. Co-existing liver diseases such as acute or chronic viral hepatitis, alcoholic liver disease, choledocholithiasis, autoimmune hepatitis, biopsy-proven non-alcoholic fatty liver disease, Wilson's disease and hemochromatosis.
4. History or presence of hepatic decompensation (e.g., variceal bleeds, encephalopathy, or poorly controlled ascites).
5. History of urolithiasis, nephritis or renal failure (clearance of creatinine < 60 ml/mn).
6. Hepatotoxic drugs use before recruiting.
7. Fuzhenghuayu anaphylaxis.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2016-01; Primary Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Rate of patients with complete biochemical response | Week 48
  Normalization of alkaline phosphatase (ALP) or decrease of ALP by more than 40% compared to the baseline.

SECONDARY OUTCOMES:
Change in liver biopsy examinations compared to the baseline. | Week 48
  Histological evolution will be checked by liver biopsy at the end of the study to compare with baseline histological status.
GLOBE scores. | Week 48
  The prognostic scores will be calculated at end of the study by GLOBE scoring system.
Change in liver stiffness status measured by magnetic resonance elastography. | Week 48
  The change of liver stiffness status at the end of the study compared to baseline checked by magnetic resonance elastography.
Change in serum alkaline phosphatase (ALP) level | Weeks 0, 4, 8, 12, 24, and 48
  Change in serum levels of ALP (IU/L) compared to the baseline.
Change in serum bilirubin level | Weeks 0, 4, 8, 12, 24, and 48
  Change in serum levels of bilirubin (mg/dL) compared to the baseline
Change in serum transaminase level | Weeks 0, 4, 8, 12, 24, and 48
  Change in serum levels of transaminase (IU/L) compared to the baseline.

OTHER OUTCOMES:
Change in pruritus from baseline | Week 48
  The symptom of pruritus will be evaluated by questionnaire before enrollment and at the end of the study.
Change in fatigue from baseline | Week 48
  The symptom of fatigue will be evaluated by Fatigue Impact Scale before enrollment and at the end of the study.
Change in serum Immunoglobulin M Levels | Week 48
  Change in serum levels of Immunoglobulin M (g/L) compared to the baseline.

CONTACTS AND LOCATIONS:
Locations (1):
- Xijing Hosipital of Digestive Disease, Xi'an, Shaanxi, China